CLINICAL TRIAL: NCT06469463
Title: Decoding Motor Imagery From Non-invasive Brain Recordings as a Prerequisite for Innovative Motor Rehabilitation Therapies
Acronym: MODECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL23_1346; 2024-A00161-46 (Other: ID-RCB)
Record Dates: First submitted 2024-05-28; First posted 2024-06-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Stroke Sequelae; Motor Imagery; Upper Limb Deficit
Keywords: Motor imagery; motor rehabilitation; magnetoencephalography; electroencephalography
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Control group of healthy subjects
  Interventions: Device: MRI; Device: MEG; Device: EEG
- Patients group (Active Comparator): Patients group of post-stroke with upper-limb deficits on one side
  Interventions: Device: EEG

INTERVENTIONS:
Device: MRI — The healthy subjects in the control group will perform an MRI head scan, which will be used to construct 3D head models and headcasts.
  Arms: Control group
Device: MEG — The healthy subjects will undergo hpMEG data while wearing 3D-printed headcasts created from high resolution MRI
  Arms: Control group
Device: EEG — The healthy participants will undergo a similar session using EEG recording, using a Polhemus Fastrak system for localization of EEG electrodes and precise co-registration with anatomy and hpMEG data.
  The patients group will take part in the same EEG recording session.

SUMMARY:
Seminal studies in motor neuroscience involving healthy subjects have revealed time-locked changes in induced power within specific frequency bands. Brain recordings were shown to exhibit a gradual reduction in signal power, relative to baseline, in the mu and beta frequency bands during an action or during motor imagery: the event-related desynchronization (ERD). This is considered to reflect processes related to movement preparation and execution and is particularly pronounced in the contralateral sensorimotor cortex. Shortly following the completion of the task, a relative increase in power, the event-related synchronization (ERS), could be observed in the beta band. ERS is thought to reflect the re-establishment of inhibition in the same area.

Ever since the characterization of the ERD and ERS phenomena, there has been little to no discussion in the field of non-invasive Brain Computer Interfaces (BCI) as to whether these features accurately capture the task-related modulations of brain activity. Recent studies in neurophysiology have demonstrated that the ERD and ERS patterns only emerge as a result of averaging signal power over multiple trials. On a single trial level, beta band activity occurs in short, transient events, bursts, rather than as sustained oscillations. This indicates that the ERD and ERS patterns reflect accumulated, time-varying changes in the burst probability during each trial. Thus, beta bursts may carry more behaviourally relevant information than averaged beta band power. Studies in humans involving arm movements have established a link between the timing of sensorimotor beta bursts and response times before movement, as well as behavioural errors post-movement. Beta burst activity in frontal areas has also been shown to correlate with movement cancellation and recent studies show that activity at the motor unit level also occurs in a transient manner, which is time-locked to sensorimotor beta bursts.

Although beta burst rate has been shown to carry significant information, it still comprises a rather simplistic representation of the underlying activity. Indeed, complex burst waveforms are embedded in the raw signals, and can be characterized by a stereotypical average shape with large variability around it. The waveform features are neglected in standard BCI approaches, because conventional signal processing methods generally presuppose sustained, oscillatory and stationary signals, and are thus inherently unsuitable for analysing transient activity.

In contrast to beta, activity in the mu frequency band is oscillatory even in single trials. This activity is typically analysed using time-frequency decomposition techniques, which assume that the underlying signal is sinusoidal. However, there is now growing consensus that oscillatory neural activity is often non-sinusoidal and that the raw waveform shape can be informative of movement.

In this project, the design of a subject-specific neurophysiological model to guide motor BCI training will be optimized using Magnetic Resonance Imaging (MRI) and Magnetoencephalography (MEG) for high spatial and biophysical specificity in the experimental group. Anatomical MR volumes will be used to design and 3D-print an individual head cast that will be used in the MEG scanner to stabilize the head position and minimize movements. This high-precision approach (hpMEG) has been proven to significantly improve source localization up to the level of distinguishing laminar activity, which makes it superior to EEG recording technique. An individualized hpMEG approach, as well as the widely adopted EEG, will be used to study bursts of oscillatory activity in the beta and mu frequency bands related to motor imagery and motor execution. hpMEG will yield subject-specific models of motor imagery that will be used to constrain online decoding of EEG data. This approach will be applied and validated on a group of healthy adult subjects and will then be compared against another feasibility group of patients and age-matched healthy participants. The proposed approach will be compared with a classic EEG-based BCI approach.

The information will be used to optimally guide subsequent EEG-based BCI training in the control group. After a thorough investigation in healthy subjects in this project, the feasibility of the approach will be evaluated in a few stroke patients with upper-limb motor deficits. Tasks 1.1 and 1.2 aim to develop subject-specific generative models decoding movement onset and offset, the type of movement, as well as finely discretized movement amplitude during both real and imagined wrist extensions/flexions. Task 1.2 investigates how lesions of patients alter our ability to decode attempted wrist movements.

DETAILED DESCRIPTION:
Seminal studies in motor neuroscience involving healthy subjects have, since a long time, revealed time-locked changes in induced power within specific frequency band. Brain recordings were shown to exhibit a gradual reduction in signal power, relative to baseline, in the mu (~ 8-12 Hz) and beta (~ 13-30 Hz) frequency bands during an action or during motor imagery (MI): the so-called event-related desynchronization (ERD). This phenomenon is considered to reflect processes related to movement preparation and execution, and is particularly pronounced in the contralateral sensorimotor cortex. Moreover, shortly following the completion of the task a relative increase in power, the event-related synchronization (ERS) (also referred to as the beta rebound), could be observed in the beta band. ERS is thought to reflect the re-establishment of inhibition in the same area.

Ever since the characterization of the ERD and ERS phenomena, there has been little to no discussion in the non-invasive BCI field as to whether these features accurately capture the task-related modulations of brain activity. Recent studies in neurophysiology have challenged this view and have demonstrated that the ERD and ERS patterns only emerge as a result of averaging signal power over multiple trials. On a single trial level, beta band activity occurs in short, transient events, termed bursts, rather than as sustained oscillations. This indicates that the ERD and ERS patterns reflect accumulated, time-varying changes in the burst probability during each trial. Thus, beta bursts may carry more behaviorally relevant information than averaged beta band power. Indeed, studies in humans involving arm movements have established a link between the timing of sensorimotor beta bursts and response times prior to movement, as well as behavioral errors post-movement. Beta burst activity in frontal areas has also been shown to correlate with movement cancellation and recent studies show that activity at the motor unit level also occurs in a transient manner, which is time-locked to sensorimotor beta bursts.

Although beta burst rate has been shown to carry significant information, it still comprises a rather simplistic representation of the underlying activity. Every burst can be characterized by a set of TF-based features: the burst peak time and peak frequency, as well as its duration and its span in the frequency axis. In turn, all these descriptors are extracted using a particular time-frequency transformation and constitute simpler representations of the more complex burst waveform that is embedded in the raw signals, and which is characterized by a stereotypical average shape with large variability around it. The waveform features are neglected in standard BCI approaches, because conventional signal processing methods generally presuppose sustained, oscillatory and stationary signals, and are thus inherently unsuitable for analyzing transient activity.

In contrast to beta, activity in the mu frequency band is oscillatory even in single trials. This activity is typically analyzed using time-frequency decomposition techniques, which assume that the underlying signal is sinusoidal. However, there is now growing consensus that oscillatory neural activity is often non-sinusoidal, and that the raw waveform shape can be informative of movement. Future efforts could take advantage of this possibility by using recently developed non-parametric cycle-by-cycle analyzes.

In this project, the investigators will optimize the design of a subject-specific neurophysiological model to guide motor BCI training, by using Magnetic Resonance Imaging (MRI) and Magnetoencephalography (MEG) for high spatial and biophysical specificity in the experimental group. Anatomical MR volumes will be used to design and 3D-print an individual head-cast that will be used in the MEG scanner in order to stabilize the subject's head position and minimize movements. This high precision approach (hpMEG) has been proven to significantly improve source localization up to the level of distinguishing laminar activity, which makes it a superior-to-EEG recording technique. In MODECO the investigators will use an individualized hpMEG approach, as well as the widely adopted EEG, to study bursts of oscillatory activity in the beta and mu frequency bands related to motor imagery and motor execution. hpMEG will yield subject-specific models of motor imagery that will be used to constrain online decoding of EEG data. This approach will be applied and validated on a group of healthy adult subjects (control group) and will then be compared against another feasibility group of patients (patient group) and age-matched healthy participants (control group; the investigators will attempt to recruit patients relatives). the investigators will compare the proposed approach with a classic EEG-based BCI approach.

the investigators will investigate how to use this information to optimally guide subsequent EEG-based BCI training in the control group. After a thorough investigation in healthy subjects in this project, the investigators will be able to evaluate this approach on a population of stroke patients with upper-limb motor deficits. Two tasks have been designed in this project tasks 1.1 and task 1.2. The aim of Task 1.1 is to develop subject-specific generative models decoding movement onset and /offset, the type of movement (left versus right), as well as finely discretized movement amplitude during both real and imagined wrist extension/flexion movements. In task 1.2 the investigators aim to investigate how the lesions of patients alter our ability to decode attempted wrist movements (control vs patients group).

ELIGIBILITY:
Inclusion Criteria:

Control group:

* Healthy subjects with age> 18, male or female.
* Right handed (Due to the fact that unlike right-handed people, left-handed people tend to have more complicated somatotopic organization of the motor cortex, we will avoid confounding observed differences to differences attributable to anatomic factors).
* Registered with the French healthcare system.
* Motivated to participate in the study.
* Normal or corrected vision.
* Adequate knowledge of French language to be able to follow directions.
* Subjects must be able to listen and understand the study instructions.
* Subjects must be able to give written informed consent before participation.
* No history of neurological or psychiatric disease.
* No physical disability of the arms or wrists.
* No use of drugs affecting the central nervous system or self-reported abuse of any drugs.

Patient group :

* Male or female stroke patients over 18 years old.
* Stroke patients must be not be in the acute phase of stroke.
* Right-handed.
* Having motor disorders in at least one of the upper limbs following the stroke, possibly with moderate accompanying deficits but no cognitive deficits.
* Entitled to a social security scheme.
* Motivated to participate in the study.
* Having normal or corrected vision.
* Having a sufficient understanding of the French language to be able to follow directions.
* Able to listen and understand study instructions.
* Able to give their written informed consent before participating.

Exclusion Criteria:

* Subjects with characteristics incompatible with MEG and MRI :

  1. Claustrophobia.
* Subjects with motor impairment (only applies to control group), severe traumatic brain injury.
* Subjects with chronic stroke (applies to both groups).
* Subjects history of skin disease or skin allergies (multiple or severe).
* Subjects who:

  1. have had an MRI within 2 weeks prior to the experiment.
  2. have implanted materials (any dental apparatus containing metal including or root canals or any metallic object, pacemaker, cochlear implanted in the body).
* Subjects working with metals in their professional lives.
* Pregnant or lactating women Pregnant or lactating women (check with a urinary test).
* Subjects who are not able to tolerate sitting for longer than 2 hours (the estimated length of an experimental session is about 2h30mins).
* Subjects with alcohol dependence (no consumption of alcohol or drugs at least 24 hours prior to the day of experiments).
* Subjects currently taking a medication that may have a strong effect on MEG or EEG recordings (e.g., antidepressants, stimulant medication, etc).
* Subjects who, in the opinion of the investigator, are not able or willing to comply with the protocol.
* Persons under guardianship or curatorship.
* Persons in emergency situations who cannot give their consent.
* Subjects under 18 years of age.
* Subjects under legal protection measures.
* Volunteers with contraindications to MEG examination
* Pacemaker.
* Implanted pump including insulin pump.
* Neurostimulator.
* Cochlear implants or other hearing aids.
* Metal prosthesis.
* Intracerebral / surgical aneurysm clips.
* Ocular or cerebral ferromagnetic foreign bodies in the upper body.
* Neurosurgical ventriculoperitoneal shunt valves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Develop subject-specific generative models | 2 years
  Movement Onset and Offset Detected During Real and Imagined Wrist Extension/Flexion Movements.
  Direction of Movement Detected During Real and Imagined Wrist Extension/Flexion Movements.
  Amplitude of Movement Measured During Real and Imagined Wrist Extension/Flexion Movements.
  Each of these outcome measures focuses on a specific aspect of the movement, providing all the necessary information to developp subject-specific generative models.

SECONDARY OUTCOMES:
Beta burst characterization. | 2 years
  Timing of Beta Bursts Measured in MEG & EEG Recordings. Location of Beta Bursts Measured in MEG & EEG Recordings. Waveform Shape of Beta Bursts Measured in MEG & EEG Recordings.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Neurosciences de Lyon - INSERM U1028, Bron, France